CLINICAL TRIAL: NCT04579757
Title: An Open-Label Phase Ib/II Study of Surufatinib in Combination With Tislelizumab in Subjects With Advanced Solid Tumors
Brief Title: Surufatinib in Combination With Tislelizumab in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Hutchmed (Industry)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-012-GLOB1
Record Dates: First submitted 2020-09-02; First posted 2020-10-08 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Solid Tumor; Colorectal Cancer; Neuroendocrine Tumors; Small Cell Lung Cancer; Gastric Cancer; Soft Tissue Sarcoma; Anaplastic Thyroid Cancer
Keywords: VEGF; PD-1
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Neuroendocrine Tumors; Small Cell Lung Carcinoma; Stomach Neoplasms; Sarcoma; Thyroid Carcinoma, Anaplastic | interventions — surufatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surufatinib and tislelizumab (dose escalation_Part 1) (Experimental): In Part 1 (dose escalation), surufatinib and will be administered orally (PO) once daily (QD) and tislelizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W).
  Interventions: Drug: Surufatinib and Tislelizumab _ Part 1
- Surufatinib and tislelizumab (indication specific_Part 2) (Experimental): In Part 2, the indication-specific expansion portion of the study, patients will receive surufatinib at the Recommended Phase 2 Dose (RP2D) dose selected in Part 1 with 200 mg tislelizumab IV, Q3W
  Interventions: Drug: Surufatinib and Tislelizumab _ Part 2

INTERVENTIONS:
Drug: Surufatinib and Tislelizumab _ Part 1 — Part 1 (all cohorts): oral surufatinib at a dose based on cohort level and intravenous tislelizumab at a 200-mg dose
  Other Names: HMPL-012, sulfatinib, BGB-A317
  Arms: Surufatinib and tislelizumab (dose escalation_Part 1)
Drug: Surufatinib and Tislelizumab _ Part 2 — Part 2 (all cohorts): oral surufatinib at the RP2D dose selected in Part 1 and intravenous tislelizumab at a 200-mg dose
  Other Names: HMPL-012, sulfatinib, BGB-A317
  Arms: Surufatinib and tislelizumab (indication specific_Part 2)

SUMMARY:
This open-label, phase Ib/II study of surufatinib in combination with tislelizumab will evaluate the safety, tolerability, PK and efficacy in patients with advanced solid tumors. The study consists of 2 parts - dose finding (Part 1) and dose expansion (Part 2).

DETAILED DESCRIPTION:
This open-label, phase Ib/II study of surufatinib in combination with tislelizumab will evaluate the safety, tolerability, PK and efficacy in patients with advanced solid tumors. The study consists of 2 parts - dose finding (Part 1) and dose expansion (Part 2).

Part 1 will be conducted to determine the recommended phase 2 dose (RP2D) and/or the maximum tolerated dose (MTD) of surufatinib in combination with tislelizumab in patients with advanced or metastatic solid tumors who have progressed on, or are intolerant to standard therapies.

Part 2 will be an open-label, multi-cohort design to evaluate the anti-tumor activity of surufatinib in combination with tislelizumab in patients with specific types of advanced or metastatic solid tumors. Patients will receive the RP2D determined in part 1 of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. ≥18 years of age
3. Part 1-have evaluable lesions (according to Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1])
4. Part 2-have measurable lesions (according to RECIST v1.1)
5. Have a performance status of 0 or 1 on the ECOG scale
6. For female subjects of childbearing potential and male patients with partners of childbearing potential, agreement to use a highly effective form(s) of contraception

   Dose Escalation:
7. Histologically or cytologically documented, locally advanced or metastatic solid malignancy of any type,.

   Dose Expansion:
8. Histologically or cytologically documented, locally advanced or metastatic:

Cohort A: adenocarcinoma of the colon or rectum that is microsatellite stable. Subjects must have progressed on, or had intolerable toxicity to, at least 3 prior regimens of standard chemotherapy.

Cohort B: progressive, low or intermediate grade (grade 1 or grade 2) NETs of thoracic or GEP origins. Subjects must have radiological documentation of progression of disease in the last 6 months and must have progressed on at least one line of standard therapy for metastatic disease.

Cohort C: SCLC that has progressed on standard first line chemotherapy treatment.

Cohort D: adenocarcinoma of the stomach or gastroesophageal junction and have progressed on at least 2 prior lines of therapy. Tumor stain for PD-L1 by Combined Positive Score (CPS) ≥5%.

Cohort E: ASPS or UPS. Subjects must have radiological documentation of disease progression in the last 3 months and have progressed on at least one line of standard therapy or refused standard frontline cytotoxic chemotherapy.

Cohort F: Anaplastic thyroid cancer that is considered not curable by resection. Patients with a BRAFV600E mutation must have previously been treated with 1 line of systemic therapy with a BRAF-targeted therapy.

Exclusion Criteria:

1. Adverse events (AEs) due to previous anti-tumor therapy has not recovered to Common Terminology Criteria for Adverse Event (CTCAE) ≤Grade 1;
2. Part 2 subjects with CRC , NETs and STS any previous treatment with anti-PD-1, anti PD-L1/L2 antibodies, anti-cytotoxic T lymphocyte associated antigen-4 (CTLA-4) antibody, or any other antibody acting on T cell costimulatory or checkpoint pathway;
3. Previous treatment with surufatinib;
4. Uncontrollable hypertension;
5. History or presence of a serious hemorrhage (>30 ml within 3 months), hemoptysis (>5 ml blood within 4 weeks) or life threatening thromboembolic event within 6 months;
6. Clinically significant cardiovascular disease;
7. Any clinically significant active infection, including, but not limited to, known human immunodeficiency virus (HIV) infection;
8. Brain metastases and/or leptomeningeal disease and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of SD for 14 days or longer; subjects requiring steroids within 4 weeks prior to start of study treatment will be excluded;
9. Active autoimmune diseases or history of autoimmune diseases that may relapse with the following exceptions:

   1. Controlled Type 1 diabetes
   2. Hypothyroidism (provided it is managed with hormone-replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, or alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors.
10. Arterial thrombosis or thromboembolic events (including stroke and/or transient ischemic attack) within 12 months prior to first dosing;
11. History of deep venous thrombosis within 6 months;
12. Female patients who are pregnant or breastfeeding;
13. Any condition by which investigators judge patients not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, MD, Study Chair — Hutchmed
Locations (18):
- United States (18):
  - Arizona Oncology Associated, PC-HOPE, Tucson, Arizona
  - City of Hope, Duarte, California
  - Rocky Mountain Cancer Centers Midtown, Denver, Colorado
  - Johns Hopkins University - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Holden Comprehensive Cancer Center, University of Iowa, Iowa City, Iowa
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Prisma Health - Upstate (ITOR), Greenville, South Carolina
  - Sarah Cannon, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 1b/2, 2-part, open-label study was conducted in patients with advanced solid tumors.
Pre-assignment Details: The study consisted of a dose-escalation phase and a dose-expansion phase. A total of 12 patients in dose-escalation phase and 75 patients in dose-expansion phase were enrolled in this study. The study was terminated early based on the strategic re-evaluation of clinical development of surufatinib in the United States and Europe with no safety concerns. No patients were enrolled in Cohort E1 (alveolar soft part sarcoma) in the dose-expansion phase, hence this cohort is not presented in results.
Groups:
- Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab: Patients with advanced or metastatic solid tumors of any kind who had progressed on or were intolerant of standard therapies received surufatinib 250 milligrams (mg) orally once daily (QD) in combination with tislelizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) until progressive disease (PD), unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab: Patients with advanced or metastatic solid tumors of any kind who had progressed on or were intolerant of standard therapies received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort A: CRC: Patients with microsatellite stable, locally advanced or metastatic colorectal cancer (CRC) that was previously treated with at least 3 prior lines of therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort B1: Thoracic NETs: Patients with thoracic neuroendocrine tumor (NET) who had progressive, locally advanced or metastatic, low-to-intermediate grade (Grade 1 or Grade 2), well-differentiated NETs that progressed on at least 1 line of standard therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort B2: GEP NETs: Patients with gastroenteropancreatic (GEP) NET who had progressive, locally advanced or metastatic, low-to-intermediate grade (Grade 1 or Grade 2), well-differentiated NETs that progressed on at least 1 line of standard therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort C: SCLC: Patients with locally advanced or metastatic small-cell lung cancer (SCLC) that was previously progressed on first-line chemotherapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort D: GC: Patients with microsatellite stable, programmed death-ligand 1 (PD-L1) ≥5%, locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction (gastric cancer [GC]), and were previously treated with at least 2 lines of standard therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort E2: UPS: Patients with undifferentiated pleomorphic sarcoma (UPS) who progressed on, or had discontinued due to intolerable toxicity to, at least 1 line of standard therapy or were unsuitable for standard frontline cytotoxic chemotherapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort F: ATC: Patients with locally advanced or metastatic anaplastic thyroid cancer (ATC) and who had a B-Raf kinase V600E (BRAFV600E) mutation were previously treated with 1 line of systemic therapy (not including radiation therapy) with a BRAF-targeted therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
Period: Overall Study
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Started | 6 | 6 | 15 | 10 | 20 | 15 | 3 | 9 | 3
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not Completed | 6 | 6 | 15 | 10 | 19 | 15 | 3 | 8 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Death | 4 | 1 | 14 | 3 | 2 | 7 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 3 | 0
Not completed — Radiological or Clinical PD | 1 | 4 | 1 | 3 | 9 | 4 | 2 | 2 | 0
Not completed — Start of New Therapy | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Groups:
- Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab: Patients with advanced or metastatic solid tumors of any kind who had progressed on or were intolerant of standard therapies received surufatinib 250 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort A: CRC: Patients with microsatellite stable, locally advanced or metastatic CRC that was previously treated with at least 3 prior lines of therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort B1: Thoracic NETs: Patients with thoracic NET who had progressive, locally advanced or metastatic, low-to-intermediate grade (Grade 1 or Grade 2), well-differentiated NETs that progressed on at least 1 line of standard therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort B2: GEP NETs: Patients with GEP NET who had progressive, locally advanced or metastatic, low-to-intermediate grade (Grade 1 or Grade 2), well-differentiated NETs that progressed on at least 1 line of standard therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort C: SCLC: Patients with locally advanced or metastatic SCLC that was previously progressed on first-line chemotherapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort D: GC: Patients with microsatellite stable, PD-L1 ≥5%, locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction (GC) and were previously treated with at least 2 lines of standard therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort E2: UPS: Patients with UPS who progressed on, or had discontinued due to intolerable toxicity to, at least 1 line of standard therapy or were unsuitable for standard frontline cytotoxic chemotherapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Dose Expansion Phase: Cohort F: ATC: Patients with locally advanced or metastatic ATC and who had a BRAFV600E mutation were previously treated with 1 line of systemic therapy (not including radiation therapy) with a BRAF-targeted therapy received surufatinib 300 mg orally QD in combination with tislelizumab 200 mg IV infusion Q3W until PD, unacceptable toxicity, withdrawal of consent, new anticancer therapy, lost to follow-up, or death.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC | Total
Number analyzed (Participants) | 6 | 6 | 15 | 10 | 20 | 15 | 3 | 9 | 3 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (14.69) | 68.2 (9.83) | 53.5 (11.99) | 58.6 (9.70) | 63.2 (9.23) | 58.1 (14.27) | 60.7 (5.86) | 59.9 (13.94) | 63.0 (19.05) | 60.0 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 8 | 4 | 10 | 8 | 0 | 6 | 1 | 40
  Male | 5 | 4 | 7 | 6 | 10 | 7 | 3 | 3 | 2 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 5 | 6 | 15 | 9 | 18 | 13 | 3 | 8 | 2 | 79
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 4 | 0 | 3 | 1 | 0 | 0 | 0 | 9
  White | 3 | 3 | 10 | 8 | 17 | 12 | 3 | 9 | 3 | 68
  More than one race | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Number of Patients With Dose-Limiting Toxicities (DLTs)
Description: According to National Cancer Institute Common Terminology Criteria for Adverse Events(AEs) version (v)5.0,DLT was defined as any of the following AEs during DLT observation period:
  Nonhematologic toxicities:grade 3 or higher nonhematologic toxicity, except for grade 3 fatigue lasting <7 days, grade 3 rash returning to baseline or ≤grade 1 within 7 days with treatment, grade 3 hypertension downgraded to ≤grade 1 within 7 days with therapy, grade 3 endocrinopathy controlled by hormonal replacement with no hospitalization and resolving to ≤grade 1 within 7 days, grade 3 or higher amylase or lipase elevation without symptoms of pancreatitis, grade 3 nausea/vomiting or diarrhea for <72 hours with care, grade 3 or higher electrolyte abnormality lasting up to 72 hours and resolving with treatment. Hematologic toxicities: grade 3 or higher febrile neutropenia, grade 4 neutropenia and grade 4 thrombocytopenia lasting >7 days, grade 3 thrombocytopenia with severe bleeding, and grade 4 anemia.
Time Frame: From the first dose of study drug (Day 1) up to Day 21 of Cycle 1 (cycle duration: 3 weeks)
Population: The DLT-evaluable analysis set included all patients enrolled in dose escalation phase of the study who were evaluable for DLT assessment and received ≥85% of scheduled surufatinib and ≥67% of scheduled tislelizumab administration during the DLT assessment window and/or experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

2. Primary Outcome: Dose Escalation Phase: Number of Patients With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and TEAEs Leading to Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a clinical study patient temporally associated with the use of a study treatment in humans, whether or not considered related to the treatment. An AE was considered "serious" if, in the view of either the investigator or sponsor, it resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, was a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that started or worsened in severity on or after the first dose of study treatment and up to 30 days after the date of last study treatment administration.
Time Frame: From the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 9 months
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab
Number analyzed (Participants) | 6 | 6
Participants
  Any TEAEs | 6 | 6
  Any TESAEs | 5 | 3
  Any TEAEs leading to surufatinib treatment discontinuation | 3 | 0
  Any TEAEs leading to tislelizumab treatment discontinuation | 3 | 0

3. Primary Outcome: Dose Expansion Phase: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of patients with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Tumor assessments performed every 6 weeks (+/-1 week) for the first 24 weeks and every 9 weeks (+/-1 week) thereafter, up to a maximum of approximately 37 months
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 15 | 10 | 20 | 15 | 3 | 9 | 3
percentage of patients | 6.7 [0.2 to 31.9] | 0 [NA to NA] — NA indicates that upper and lower limits of confidence interval (CI) were not estimable as there were no patients with CR or PR in that disease cohort. | 15.0 [3.2 to 37.9] | 13.3 [1.7 to 40.5] | 33.3 [0.8 to 90.6] | 44.4 [13.7 to 78.8] | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable as there were no patients with CR or PR in that disease cohort.

4. Secondary Outcome: Dose Escalation Phase: Objective Response Rate
Description: ORR was defined as the percentage of patients with a confirmed BOR of CR or PR as determined by the investigator using RECIST v1.1. BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Tumor assessments performed every 6 weeks (+/-1 week) for the first 24 weeks and every 9 weeks (+/-1 week) thereafter, up to a maximum of approximately 42 months
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab
Number analyzed (Participants) | 6 | 6
percentage of patients | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable as there were no patients with CR or PR in that disease cohort. | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable as there were no patients with CR or PR in that disease cohort.

5. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Progression-free Survival (PFS)
Description: PFS was defined as the time from the start of study treatment until the first radiographic documentation of objective progression as assessed by the investigator using RECIST v1.1, or death from any cause. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 4
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 6 | 6 | 15 | 10 | 20 | 15 | 3 | 9 | 3
months | 1.5 [1.2 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 6.0 [1.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 4.7 [2.7 to 5.4] | 4.5 [0.3 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 7.4 [3.1 to 20.0] | 1.4 [1.0 to 4.0] | 9.6 [5.6 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [1.3 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 2.8 [1.2 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure.

6. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of patients with a BOR of CR, PR, or stable disease (SD) lasting for at least 7 weeks as determined by the investigator using RECIST v1.1. BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: as for outcome 4
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 6 | 6 | 15 | 10 | 20 | 15 | 3 | 9 | 3
percentage of patients | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to no patients with CR, PR, or SD for at least 7 weeks. | 66.7 [22.3 to 95.7] | 66.7 [38.4 to 88.2] | 50.0 [18.7 to 81.3] | 70.0 [45.7 to 88.1] | 26.7 [7.8 to 55.1] | 66.7 [9.4 to 99.2] | 55.6 [21.2 to 86.3] | 33.3 [0.8 to 90.6]

7. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of patients with a BOR of CR, PR, or durable SD as determined by the investigator using RECIST v1.1. Durable SD was SD for at least 6 months. BOR was defined as the best response recorded from the start of study treatment until documented RECIST v1.1 progression or the start date of new anticancer therapy, whichever came first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: as for outcome 4
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 6 | 6 | 15 | 10 | 20 | 15 | 3 | 9 | 3
percentage of patients | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to no patients with CR, PR, or SD lasting for at least 6 months. | 50.0 [11.8 to 88.2] | 20.0 [4.3 to 48.1] | 20.0 [2.5 to 55.6] | 40.0 [19.1 to 63.9] | 13.3 [1.7 to 40.5] | 33.3 [0.8 to 90.6] | 44.4 [13.7 to 78.8] | 0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to no patients with CR, PR, or SD lasting for at least 6 months.

8. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Duration of Response (DoR)
Description: DoR was defined as the time from the first occurrence of PR or CR by RECIST v1.1, until PD or death, whichever came first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 4
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab. Only those patients with PR or CR (responders) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 4 | 0
months |  |  | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. |  | NA [15.0 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 8.3 [5.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 11.0 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. |

9. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Time to Response (TTR)
Description: TTR was defined as the time from start of study treatment until the date of first documented objective response, either CR or PR (whichever status was recorded first), according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 4 | 0
months |  |  | 2.7 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. |  | 3.9 [2.7 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 3.5 [1.3 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 2.7 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | 1.4 [1.2 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. |

10. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Plasma Concentration of Surufatinib
Description: Blood samples were collected at the specified timepoints to determine plasma concentration of surufatinib.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 5, 9, 17 and on Days 8 and 15 of Cycle 1; 2 to 4 hours post-dose on Days 1 and 15 of Cycle 1 (cycle duration: 3 weeks)
Population: The pharmacokinetic (PK) analysis set included all patients with at least 1 quantifiable concentration of surufatinib or tislelizumab. Only patients with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 6 | 6 | 15 | 10 | 19 | 15 | 3 | 9 | 2
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: Pre-dose: number analyzed (Participants) | 5 | 6 | 15 | 10 | 19 | 15 | 3 | 9 | 2
  Cycle 1 Day 1: Pre-dose | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL.
  Cycle 1 Day 1: 2 to 4 hours post-dose | 293.03 (244.593) | 576.00 (415.108) | 426.62 (312.209) | 276.36 (243.080) | 294.13 (292.335) | 406.97 (212.791) | 506.27 (653.616) | 275.64 (165.937) | 782.50 (463.155)
  Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 4 | 6 | 12 | 5 | 14 | 9 | 2 | 6 | 1
  Cycle 1 Day 8: Pre-dose | 77.00 (44.023) | 189.93 (113.750) | 170.33 (131.533) | 100.12 (71.600) | 92.26 (63.901) | 122.80 (70.875) | 109.10 (18.243) | 97.70 (40.471) | 709.00 (NA) — NA indicates that SD was not estimable for 1 patient.
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 5 | 5 | 11 | 4 | 15 | 10 | 2 | 6 | 0
  Cycle 1 Day 15: Pre-dose | 64.36 (15.246) | 181.56 (125.156) | 135.96 (83.673) | 159.00 (139.802) | 84.95 (70.121) | 96.79 (43.933) | 111.05 (19.728) | 118.92 (75.457) |
  Cycle 1 Day 15: 2 to 4 hours post-dose: number analyzed (Participants) | 3 | 3 | 13 | 4 | 12 | 11 | 2 | 7 | 0
  Cycle 1 Day 15: 2 to 4 hours post-dose | 318.67 (146.770) | 757.33 (498.399) | 657.54 (369.146) | 354.25 (52.519) | 471.78 (330.598) | 425.75 (235.698) | 188.00 (41.012) | 518.00 (302.182) |
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 5 | 4 | 10 | 3 | 9 | 11 | 2 | 2 | 1
  Cycle 2 Day 1: Pre-dose | 45.82 (27.567) | 96.80 (38.895) | 151.44 (99.521) | 89.37 (53.475) | 75.94 (53.028) | 117.68 (79.721) | 146.50 (26.163) | 71.95 (9.405) | 147.00 (NA) — NA indicates that SD was not estimable for 1 patient.
  Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 0 | 2 | 3 | 1 | 4 | 2 | 0 | 0 | 0
  Cycle 5 Day 1: Pre-dose |  | 55.25 (8.132) | 141.20 (117.885) | 41.00 (NA) — NA indicates that SD was not estimable for 1 patient. | 61.08 (22.279) | 105.70 (54.164) |  |  |
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Cycle 9 Day 1: Pre-dose |  | 65.90 (NA) — NA indicates that SD was not estimable for 1 patient. |  |  | 87.20 (14.964) | 41.70 (NA) — NA indicates that SD was not estimable for 1 patient. |  |  |
  Cycle 17 Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 17 Day 1: Pre-dose |  |  |  |  | 85.10 (NA) — NA indicates that SD was not estimable for 1 patient. |  |  |  |

11. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Serum Concentration of Tislelizumab
Description: Blood samples were collected at the specified timepoints to determine serum concentration of tislelizumab.
Time Frame: Preinfusion on Day 1 of Cycles 1, 2, 5, 9, 17; end of infusion on Day 1 of Cycles 1 and 5; on Days 8 and 15 of Cycle 1 (cycle duration: 3 weeks)
Population: The PK analysis set included all patients with at least 1 quantifiable concentration of surufatinib or tislelizumab. Only patients with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 6 | 6 | 15 | 10 | 19 | 15 | 3 | 9 | 2
ng/mL
  Cycle 1 Day 1: Preinfusion: number analyzed (Participants) | 6 | 6 | 15 | 9 | 19 | 15 | 3 | 9 | 2
  Cycle 1 Day 1: Preinfusion | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 400 ng/mL.
  Cycle 1 Day 1: End of Infusion | 44550.0 (7420.98) | 62750.0 (17420.53) | 57233.3 (8846.28) | 70990.0 (41600.73) | 61136.8 (15927.90) | 66220.0 (17336.43) | 67966.7 (45015.59) | 55955.6 (15499.61) | 42200.0 (12727.92)
  Cycle 1 Day 8: number analyzed (Participants) | 6 | 6 | 13 | 8 | 18 | 12 | 3 | 8 | 2
  Cycle 1 Day 8 | 16980.0 (6850.75) | 26216.7 (7702.32) | 26446.2 (6387.83) | 29575.0 (5751.46) | 32244.4 (7253.58) | 35450.0 (8899.39) | 38233.3 (35800.33) | 25475.0 (6549.10) | 16050.0 (1767.77)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 6 | 12 | 7 | 16 | 12 | 2 | 8 | 2
  Cycle 1 Day 15 | 14296.7 (5945.36) | 17900.0 (5297.55) | 17414.2 (4199.94) | 20571.4 (2817.63) | 24506.3 (6403.07) | 23783.3 (4274.20) | 43950.0 (40658.64) | 19300.0 (4755.45) | 10940.0 (2489.02)
  Cycle 2 Day 1: Preinfusion: number analyzed (Participants) | 5 | 5 | 14 | 6 | 15 | 12 | 2 | 8 | 2
  Cycle 2 Day 1: Preinfusion | 9564.0 (7871.14) | 13804.0 (4782.16) | 13858.6 (4730.49) | 14033.3 (2436.12) | 18020.0 (5688.23) | 17725.0 (3860.55) | 38000.0 (36910.97) | 12161.3 (4443.93) | 7640.0 (2729.43)
  Cycle 5 Day 1: Preinfusion: number analyzed (Participants) | 0 | 3 | 8 | 1 | 8 | 4 | 1 | 3 | 1
  Cycle 5 Day 1: Preinfusion |  | 24400.0 (14028.90) | 36412.5 (34947.57) | 46400.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 41575.0 (10065.32) | 31225.0 (12388.81) | 20100.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 19200.0 (3143.25) | 22700.0 (NA) — NA indicates that SD was not estimable for 1 patient.
  Cycle 5 Day 1: End of Infusion: number analyzed (Participants) | 0 | 3 | 7 | 2 | 8 | 4 | 1 | 3 | 1
  Cycle 5 Day 1: End of Infusion |  | 87166.7 (34425.04) | 102500.0 (26662.02) | 117500.0 (6363.96) | 113475.0 (16286.34) | 117550.0 (43800.65) | 80800.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 103033.3 (17737.06) | 69000.0 (NA) — NA indicates that SD was not estimable for 1 patient.
  Cycle 9 Day 1: Preinfusion: number analyzed (Participants) | 0 | 2 | 1 | 1 | 5 | 2 | 0 | 2 | 0
  Cycle 9 Day 1: Preinfusion |  | 22700.0 (4101.22) | 44800.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 50000.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 45500.0 (5384.24) | 41200.0 (24607.32) |  | 41100.0 (16970.56) |
  Cycle 17 Day 1: Preinfusion: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0
  Cycle 17 Day 1: Preinfusion |  |  |  | 41300.0 (NA) — NA indicates that SD was not estimable for 1 patient. | 44766.7 (12196.86) | 51900.0 (NA) — NA indicates that SD was not estimable for 1 patient. |  | 47300.0 (NA) — NA indicates that SD was not estimable for 1 patient. |

12. Secondary Outcome: Dose Escalation and Dose Expansion Phases: Number of Patients With Antidrug Antibodies (ADA) to Tislelizumab
Description: Blood samples were collected at the specified timepoints to detect ADAs to tislelizumab. Treatment-boosted ADA was defined as ADA positive at baseline that was boosted to a 4-fold or higher-level following treatment administration. Treatment-induced ADA was defined as ADA negative at baseline and ADA positive post-baseline.
Time Frame: From the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 9 months for dose escalation phase and approximately 33 months for dose expansion phase
Population: The ADA analysis set included all patients who received at least 1 dose of tislelizumab and had a baseline and at least 1 post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 6 | 5 | 14 | 8 | 16 | 13 | 2 | 9 | 2
Participants
  Treatment-Boosted ADA | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-Induced ADA | 2 | 2 | 5 | 3 | 5 | 1 | 0 | 5 | 1

13. Secondary Outcome: Dose Expansion Phase (Cohorts A and F): Overall Survival (OS)
Description: OS was defined as the time from the start of study treatment until the date of death due to any cause.
Time Frame: From the first dose of study treatment (Day 1) up to date of death due to any cause, up to approximately 42 months
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab. As pre-specified in the protocol and statistical analysis plan (SAP), OS was assessed only in Cohort A (CRC) and Cohort F (ATC) of the dose expansion phase.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 15 | 3
months | 7.1 [4.8 to 11.8] | 5.3 [2.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure.

14. Secondary Outcome: Dose Expansion Phase: Number of Patients With Treatment-Emergent Adverse Events, Treatment-Emergent Serious Adverse Events and TEAEs Leading to Treatment Discontinuation
Description: as for outcome 2
Time Frame: From the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 33 months
Population: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
Number analyzed (Participants) | 15 | 10 | 20 | 15 | 3 | 9 | 3
Participants
  Any TEAEs | 14 | 10 | 20 | 15 | 3 | 9 | 3
  Any TESAEs | 9 | 5 | 9 | 8 | 0 | 4 | 1
  Any TEAEs leading to surufatinib treatment discontinuation | 3 | 2 | 5 | 5 | 0 | 2 | 0
  Any TEAEs leading to tislelizumab treatment discontinuation | 6 | 2 | 6 | 5 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 9 months for dose escalation phase and approximately 33 months for dose expansion phase. All-cause mortality (deaths) were collected from signing of the informed consent form up to end of follow up, approximately 42 months.
Description: The SAS included all enrolled patients who received at least 1 dose of surufatinib or tislelizumab.
Arm/Group | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab | Dose Expansion Phase: Cohort A: CRC | Dose Expansion Phase: Cohort B1: Thoracic NETs | Dose Expansion Phase: Cohort B2: GEP NETs | Dose Expansion Phase: Cohort C: SCLC | Dose Expansion Phase: Cohort D: GC | Dose Expansion Phase: Cohort E2: UPS | Dose Expansion Phase: Cohort F: ATC
All-Cause Mortality (participants affected / at risk) | 4/6 | 1/6 | 14/15 | 4/10 | 2/20 | 8/15 | 0/3 | 1/9 | 3/3
Serious Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 9/15 | 5/10 | 9/20 | 8/15 | 0/3 | 4/9 | 1/3
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 14/15 | 10/10 | 20/20 | 15/15 | 3/3 | 8/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab (N=6) | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab (N=6) | Dose Expansion Phase: Cohort A: CRC (N=15) | Dose Expansion Phase: Cohort B1: Thoracic NETs (N=10) | Dose Expansion Phase: Cohort B2: GEP NETs (N=20) | Dose Expansion Phase: Cohort C: SCLC (N=15) | Dose Expansion Phase: Cohort D: GC (N=3) | Dose Expansion Phase: Cohort E2: UPS (N=9) | Dose Expansion Phase: Cohort F: ATC (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase: Surufatinib 250 mg + Tislelizumab (N=6) | Dose Escalation Phase: Surufatinib 300 mg + Tislelizumab (N=6) | Dose Expansion Phase: Cohort A: CRC (N=15) | Dose Expansion Phase: Cohort B1: Thoracic NETs (N=10) | Dose Expansion Phase: Cohort B2: GEP NETs (N=20) | Dose Expansion Phase: Cohort C: SCLC (N=15) | Dose Expansion Phase: Cohort D: GC (N=3) | Dose Expansion Phase: Cohort E2: UPS (N=9) | Dose Expansion Phase: Cohort F: ATC (N=3)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 10 (18) | 5 (10) | 12 (17) | 6 (12) | 3 (4) | 4 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 6 (14) | 3 (15) | 11 (19) | 6 (8) | 3 (7) | 4 (16) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 7 (13) | 3 (4) | 6 (10) | 4 (6) | 0 (0) | 3 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 3 (4) | 4 (8) | 4 (6) | 5 (5) | 2 (3) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (4) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (5) | 6 (9) | 5 (11) | 11 (14) | 7 (8) | 3 (4) | 4 (6) | 1 (2)
Oedema peripheral (General disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (2) | 7 (12) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 9 (9) | 4 (10) | 11 (13) | 3 (3) | 3 (3) | 3 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (8) | 2 (2) | 5 (8) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (36) | 3 (7) | 0 (0) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (6) | 3 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (8) | 5 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 4 (7) | 3 (11) | 13 (37) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 2 (9) | 11 (26) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 5 (7) | 2 (2) | 7 (24) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 1 (1) | 4 (4) | 4 (5) | 2 (7) | 3 (3) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 3 (5) | 2 (5) | 6 (12) | 1 (3) | 1 (1) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (6) | 5 (16) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 4 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (14) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 10 (23) | 3 (7) | 9 (37) | 1 (1) | 1 (4) | 4 (8) | 2 (4)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 6 (7) | 4 (4) | 0 (0) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 5 (7) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 3 (3) | 2 (2) | 0 (0) | 3 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 8 (24) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (6) | 5 (13) | 4 (5) | 9 (47) | 0 (0) | 1 (1) | 1 (10) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (3) | 1 (1) | 3 (3) | 4 (11) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on the strategic re-evaluation of the clinical development of surufatinib in the United States and Europe with no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04579757/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT04579757/SAP_001.pdf